CLINICAL TRIAL: NCT04841694
Title: Prospective Randomized Double-Blind Placebo Controlled Study of Oral Probiotics on the Shift of Gut Microbiome and Skin Carotenoid Levels
Brief Title: Oral Probiotics on the Shift in Gut Microbiome and Skin Carotenoid Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Microbiome labs (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, Principal Investigator, Integrative Skin Science and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROB-CAROT
Record Dates: First submitted 2021-04-05; First posted 2021-04-12 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Human Microbiome
Keywords: gut microbiome; dermatology; skin; carotenoids; probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Participants will be taking a probiotic supplement that they will be taking by mouth once per day
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Bacillus indicus

SUMMARY:
The purpose of this study is to determine how probiotics affects circulating carotenoid levels.

DETAILED DESCRIPTION:
Certain probiotic strains are rich in the production of carotenoids. This study will evaluate if probiotic supplementation with a carotenoid rich strain will augment circulating carotenoids.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 40+
* Must be willing to comply with all protocol requirements
* Must be willing to have flash photo facial images taken with the imaging systems
* Fitzpatrick skin type II, III, or IV

Exclusion Criteria:

* Any systemic or antibiotics (injected or oral) within 6 months of starting study
* Any topical antibiotic or Vitamin A within 1 month of starting study or any subject unwilling to refrain from washout of topical antibacterial or vitamin A ingredient.
* Any oral probiotic or prebiotic supplementation within past 1 month at the discretion of the investigator.
* Limit total fruit and vegetable intake to 2.5 servings (1 serving=1 cup) per day of high carotenoid foods. High carotenoid foods include spinach, summer squash, carrots, citrus fruits, celery, kale, tomatoes, and cantaloupe
* Subjects must have no history of malignancy or cancer (excluding skin cancer unless there is a history of metastasis) or diagnosis of gastrointestinal inflammatory diseases, no history or diagnosis of epilepsy, no history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis)
* Has a condition or is on medication the investigator and/or designee believe could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results
* Women who have been pregnant in the last three months, are pregnant, preparing to be pregnant or lactating.
* Is participating in a concurrent intervention based clinical research study
* Those with BMI higher than 35 kg/m²
* Commencement of a new diet (such as the ketogenic diet) or supplements within the 1 month prior to initiating participation, at the discretion of the investigator.
* Is participating in or has participated in a intervention based facial study at this or any other facility in the past 2 weeks. Participation in survey-based studies are approved at the discretion of the investigator.
* Has a skin disease on face that will interfere with image collection and assessment in the opinion of the investigator
* Refusal to shave or remove facial hair that may interfere with image collection and assessment.
* Persons unwilling to avoid the following during the 4 weeks prior and during the duration of the study: self-tanning, spa tanning, sun tanning, or artificial tanning.
* Known allergy or irritation to the supplement utilized in the study
* Persons unwilling to avoid sun exposure to the inner forearm
* Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco
* Cutaneous photosensitivity at wavelengths of 400-450 nm
* Porphyria or known allergies to porphyrins
* Prisoners
* Adults unable to consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Carotenoid Levels | 5 weeks
  Change in skin carotenoid level and blood carotenoid level with supplementation

SECONDARY OUTCOMES:
Gut Microbiome Changes | Week 5
  Shift in gut microbiome diversity
Assessment of GI related gas and constipation | Week 5
  self assessment using digestive health questionnaire
Assessment of GI related gas and constipation | Week 6
  self assessment using digestive health questionnaire
Shift in facial redness- image based | Week 5
  BTBP Clarity Mini 3D camera
Shift in facial redness- image based | Week 6
  BTBP Clarity Mini 3D camera
Shift in facial pigmentation - image based | Week 5
  BTBP Clarity Mini 3D camera
Shift in facial pigmentation - image based | Week 6
  BTBP Clarity Mini 3D camera
Protection against blue light exposure induced change in skin color | Weeks 5
  Change in skin color measured by a skin colorimeter
Protection against blue light exposure induced change in skin color | Weeks 6
  Change in skin color measured by a skin colorimeter
Carotenoid Levels | 5 weeks
  Change in skin carotenoid level and blood carotenoid level with supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No